CLINICAL TRIAL: NCT00938938
Title: Testing the Effect of Press Guides on Health Journalists
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Lisa M. Schwartz, MD, MS, White River Junction VAMC
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 16782; NCI R01CA104721
Record Dates: First submitted 2009-06-17; First posted 2009-07-14 (Estimated); Last update posted 2010-04-21 (Estimated); Status verified 2010-04

CONDITIONS: Medical Reporting
Keywords: risk communication; medical reporting; Mass media

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Press guide plus press release (Experimental): Participants in the intervention group will receive a press guide (a one-page summary of study findings written by the investigators) in addition to the journal's full narrative press release for the selected article, a copy of the article's abstract, and a link to the full text of the journal article.
  Interventions: Other: Press Guide
- Press release only (No Intervention): Participants in the control group will receive the journal's full narrative press release for the selected article, a copy of the article's abstract, and a link to the full text of the journal article.

INTERVENTIONS:
Other: Press Guide — The press guide is a 1-page summary of the study findings, written by the investigators.
  Arms: Press guide plus press release

SUMMARY:
The purpose of this study is to test the effect of adding a "press guide" to standard materials that journalists routinely receive regarding research published in medical journals.

DETAILED DESCRIPTION:
The news media has a powerful influence on public perceptions about health and health care; and much of what people -- including many physicians -- know and believe about medicine comes from the print and broadcast media. Several studies, however, have raised questions about how well the press covers medical issues, pointing out errors and omissions in coverage and misleading presentations of statistics. The goal is to help train journalists to better understand and cover medical research, and to help improve communication between journalists and medical journals.

Journalists traditionally write newspaper articles about medical research using information from press releases and the medical journal article's abstract or full text. The objective is to test whether the addition of a 'press guide' (a one-page summary of the study findings) in addition to these other materials improves comprehension of facts about the study article and the overall judgment of the newsworthiness of the study.

ELIGIBILITY:
Inclusion Criteria:

* All journalists attending the 2009 NIH/Dartmouth/VA Medicine in the Media Symposium will be invited to participate in the study.
* The symposium, which is held annually, is open to journalists across the country and from abroad.

Participants who are Health Journalists at the Health Journalism 2010 conference will be invited to participate in the study. This annual conference is being held in Chicago, IL at the Hyatt Regency McCormick Place During April 22, 2010-April 25, 2010.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Comprehension of facts about the study article (covering study design, exposures, outcome measures, results, limitations, conflicts of interest) assessed using a brief test. | 0 weeks (assessed during intervention)

SECONDARY OUTCOMES:
Overall judgment of study newsworthiness (e.g., would you argue for/against covering story with editor, how convinced are you of study validity, what headline would you write,and usefulness of press release and (intervention group) press guide. | 0 weeks (assessed during intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M. Schwartz, MD, MS, Principal Investigator — White River Junction Veterans Affairs Medical Center

REFERENCES:
- [Background] Woloshin S, Schwartz LM, Casella SL, Kennedy AT, Larson RJ. Press releases by academic medical centers: not so academic? Ann Intern Med. 2009 May 5;150(9):613-8. doi: 10.7326/0003-4819-150-9-200905050-00007. PMID 19414840